CLINICAL TRIAL: NCT06468306
Title: Combined Molecular and Mechanistic Methods for Early Detection and Individual Prevention of Pressure Ulcer Formation in Vulnerable Patients
Brief Title: Combined Molecular and Mechanistic Methods for Detection of Pressure Ulcers
Status: Not yet recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Collaborators: Region Östergötland (Other)
Responsible Party: Principal Investigator, Sara Bergstrand, Senior Associate Professor, Linkoeping University
Other Study IDs: 2023-07341-01
Record Dates: First submitted 2024-06-04; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Pressure Ulcer; Inflammatory Response
Keywords: Pressure Ulcer; nursing; prevention
MeSH Terms: conditions — Pressure Ulcer | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — skin sebum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- individuals with NIV treatment: Patients that use oronasal face masks in their ordinary care to measure early-stage medical devise-related tissue damage during routine management regimes of NIV. Approximately 150 adult patients of both sexes will be recruited, from facilities that employ oronasal face masks in the routine care.
  Interventions: Procedure: non-invasive ventilation teraphy, NIV

INTERVENTIONS:
Procedure: non-invasive ventilation teraphy, NIV — Routine management regimes of NIV

SUMMARY:
This project aims to develop a novel method for identifying early tissue damage related to pressure ulcer (PU) development in vulnerable patients by measuring biomarkers of inflammation on the skin surface. PUs are common and costly injuries that result from prolonged pressure on the skin. Current methods to assess PU risk are unreliable, and the mechanisms of PU development are not well understood. This project contributes to new knowledge of PU etiology as well as the individual variability at a molecular level combined with new knowledge about nursing actions and clinical factors linked to PU progression and outcomes of prevention. The project will use non-invasive techniques and model-based analysis to identify specific biomolecules that reflect individual susceptibility to pressure exposure in different PU risk scenarios.

DETAILED DESCRIPTION:
Purpose and aims A pressure ulcer (PU) is a localized injury to the skin and/or underlying tissue and develop from prolonged pressure on the skin. Such injuries are common in the healthcare setting, especially among vulnerable elderly. PUs greatly decrease the quality of life of individuals and are costly for the healthcare system. As many as 14% of the inpatients suffered from PUs in the Swedish country's municipalities and regions during 2022. The origin and timing of events leading to PUs are not fully understood, and current methods to assess the risk for an individual to develop a PU, are unreliable. Therefore, there is an urgent need to develop more objective, sensitive and specific methods for identifying early signs of tissue damage before they come visible and thus avoid development of PUs.

The investigators have previously identified a preliminary set of molecular biomarkers (cytokines and proteins), sampled non-invasively in the sebum, that reflects the inflammatory process under-pinning PU etiology and, possibly, individual susceptibility to pressure exposure. Therefore, it is hypothesize that non-invasive measurements of specific biomolecules on the skin surface, together with model-based analysis, can be used for individualized PU prediction. Accordingly, the purpose of this project is to confirm and expand on these preliminary findings in different PU risk scenarios to model the underlying inflammatory processes that reflect the individual vulnerability of the skin caused by pressure exposure and use modeling to extract a new layer of mechanistic insights of the underlying inflammatory process in different patient populations.

The specific aims of the project are:

1. To establish and validate optimal combinations of molecular biomarkers to identify individual susceptibility to pressure exposure during routine management regimes related to medical devises non-invasive ventilation (NIV) therapy.
2. To unravel key mechanisms in inflammatory processes related to early tissue damage by developing a mathematical model for the timing of events in the response to pressure, based on collected biomolecules, earlier data, and interaction databases
3. To identify risk factors of PU vulnerability on an individual level in routine clinical settings by combining biomolecules, model-based simulations, and clinical parameters

ELIGIBILITY:
Inclusion Criteria:

- patients that use oronasal face masks in their ordinary care during routine management regimes of non invasive ventilation.

Exclusion Criteria

* acute respiratory failure
* previous ICU care
* pressure ulcer on measurement site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that use oronasal face masks in their ordinary care during routine management regimes of non invasive ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
CTACK | 2 minutes
  inflammatory biomarker
ENA-78 | 2 minutes
  inflammatory biomarker
Eotaxin | 2 minutes
  inflammatory biomarker
Eotaxin-2 | 2 minutes
  inflammatory biomarker
Eotaxin-3 | 2 minutes
  inflammatory biomarker
EPO | 2 minutes
  inflammatory biomarker
FLT3L | 2 minutes
  inflammatory biomarker
Fractalkine | 2 minutes
  inflammatory biomarker
G-CSF | 2 minutes
  inflammatory biomarker
GM-CSF | 2 minutes
  inflammatory biomarker
GRO-alpha | 2 minutes
  inflammatory biomarker
I-309 | 2 minutes
  inflammatory biomarker
IFN-α2a | 2 minutes
  inflammatory biomarker
IFN-β | 2 minutes
  inflammatory biomarker
IFN-γ | 2 minutes
  inflammatory biomarker
IL-10 | 2 minutes
  inflammatory biomarker
IL-12/IL-23p40 | 2 minutes
  inflammatory biomarker
IL-12p70 | 2 minutes
  inflammatory biomarker
IL-13 | 2 minutes
  inflammatory biomarker
IL-15 | 2 minutes
  inflammatory biomarker
IL-16 | 2 minutes
  inflammatory biomarker
IL-17A | 2 minutes
  inflammatory biomarker
IL-17A/F | 2 minutes
  inflammatory biomarker
IL-17B | 2 minutes
  inflammatory biomarker
IL-17C | 2 minutes
  inflammatory biomarker
IL-17D | 2 minutes
  inflammatory biomarker
IL-17E/IL-25 | 2 minutes
  inflammatory biomarker
IL-17F | 2 minutes
  inflammatory biomarker
IL-18 | 2 minutes
  inflammatory biomarker
IL-1RA | 2 minutes
  inflammatory biomarker
IL-1α | 2 minutes
  inflammatory biomarker
IL-1β | 2 minutes
  inflammatory biomarker
IL-2 | 2 minutes
  inflammatory biomarker
IL-21 | 2 minutes
  inflammatory biomarker
IL-22 | 2 minutes
  inflammatory biomarker
IL-23 | 2 minutes
  inflammatory biomarker
IL-27 | 2 minutes
  inflammatory biomarker
IL-29/IFN-L1 | 2 minutes
  inflammatory biomarker
IL-2Ra | 2 minutes
  inflammatory biomarker
IL-3 | 2 minutes
  inflammatory biomarker
IL-31 | 2 minutes
  inflammatory biomarker
IL-33 | 2 minutes
  inflammatory biomarker
IL-4 | 2 minutes
  inflammatory biomarker
IL-5 | 2 minutes
  inflammatory biomarker
IL-6 | 2 minutes
  inflammatory biomarker
IL-7 | 2 minutes
  inflammatory biomarker
IL-8 | 2 minutes
  inflammatory biomarker
IL-9 | 2 minutes
  inflammatory biomarker
IP-10 | 2 minutes
  inflammatory biomarker
I-TAC | 2 minutes
  inflammatory biomarker
MCP-1 | 2 minutes
  inflammatory biomarker
MCP-2 | 2 minutes
  inflammatory biomarker
MCP-3 | 2 minutes
  inflammatory biomarker
MCP-4 | 2 minutes
  inflammatory biomarker
M-CSF | 2 minutes
  inflammatory biomarker
MDC | 2 minutes
  inflammatory biomarker
MIF | 2 minutes
  inflammatory biomarker
MIP-1α | 2 minutes
  inflammatory biomarker
MIP-1β | 2 minutes
  inflammatory biomarker
MIP-3α | 2 minutes
  inflammatory biomarker
MIP-3β | 2 minutes
  inflammatory biomarker
MIP-5 | 2 minutes
  inflammatory biomarker
SDF-1alpha | 2 minutes
  inflammatory biomarker
TARC | 2 minutes
  inflammatory biomarker
TNF-α | 2 minutes
  inflammatory biomarker
TNF-β | 2 minutes
  inflammatory biomarker
TPO | 2 minutes
  inflammatory biomarker
TRAIL | 2 minutes
  inflammatory biomarker
TSLP | 2 minutes
  inflammatory biomarker
VEGF-A | 2 minutes
  inflammatory biomarker
YKL-40 | 2 minutes
  inflammatory biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Sara Bergstrand, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linköping University, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No
No IDP data will be shared outside the research group

REFERENCES:
- [Background] Kallman U, Bergstrand S, Ek AC, Engstrom M, Lindgren M. Blood flow responses over sacrum in nursing home residents during one hour bed rest. Microcirculation. 2016 Oct;23(7):530-539. doi: 10.1111/micc.12303. PMID 27534925
- [Background] Feldt A, Kohler AK, Bergstrand S. Nurses' strategies to enable continuous positive airway pressure therapy in a general medical ward context: A qualitative study. Scand J Caring Sci. 2023 Jun;37(2):524-533. doi: 10.1111/scs.13136. Epub 2022 Nov 28. PMID 36440591
- [Background] John AJUK, Galdo FD, Gush R, Worsley PR. An evaluation of mechanical and biophysical skin parameters at different body locations. Skin Res Technol. 2023 Feb;29(2):e13292. doi: 10.1111/srt.13292. PMID 36823505
- [Background] Jayabal H, Bader DL, Worsley P. Development of an Efficient Extraction Methodology to Analyse Potential Inflammatory Biomarkers from Sebum. Skin Pharmacol Physiol. 2023;36(1):38-50. doi: 10.1159/000528653. Epub 2022 Dec 26. PMID 36572004